CLINICAL TRIAL: NCT00539825
Title: A Randomized Double-blind, Placebo-controlled, Crossover, Dose Escalation Study to Examine the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK704838 and Tiotropium Bromide
Brief Title: Effect of GSK704838 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AC6108697
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Anticholinergic,; Plethysmography; Muscarinic Receptor Antagonist,; COPD,; FTIH,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK704838

SUMMARY:
GSK704838C is a potent, pan-active mAChR antagonist, which is being developed for once-daily treatment of chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Aged between 18-55 years inclusive.
* Non-smokers
* Normal spirometry
* A signed and dated written informed consent is obtained from the subject.
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete the study.
* The subject is =50kg with a body mass index within the range 19.0 to 29.9 kg/m2 inclusive.
* Response to ipratropium bromide

Exclusion Criteria:

* Any clinically relevant and important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead or Holter).
* A history of breathing problems
* A mean QTc(B) value > 450ms, the QTc(B) of the 3 screening ECGs are not within 10% of the mean, a PR interval outside the range 90-210ms or an ECG that is not suitable for QT measurements at screening.
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 40-90 bpm inclusive at screening.
* History of use of tobacco- or nicotine-containing products within 6 months of screening, and/or positive urine cotinine test results at screening.
* Where participation in the study would result in donation of blood in excess of 500mL within a 56 day period at screening.
* The subject is currently taking regular (or a course of) medication, whether prescribed or not, including herbal remedies such as St John's Wort etc.

The subject has taken:

* prescription medications for 14 days prior to first dose of study drug, or
* Over-the-counter (OTC) medications/preparations (including herbal remedies, etc.) excluding simple analgesics for 48 hours prior to first dose of study drug, unless it is judged by the Investigator not to compromise the subject's safety or influence the outcome of the study.

  * The subject has participated in a study with a new molecular entity or any other trial within a period of 3 months prior first dose of study drug.
  * The subject has tested positive for hepatitis C antibody (third generation enzyme immunoassay), hepatitis B surface antigen or HIV antibodies (if tested according to site SOP's) at screening.
  * The subject has tested positive for drugs-of-abuse at screening.
  * The subject has tested positive for urine alcohol (including ethanol) at screening.

The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.

* The subject is unable to use the DISKUS™ and/or HandiHaler inhaler devices correctly at screening.
* The subject has a suspected history of alcohol abuse within the six months previous to the screening visit.
* The subject has a known allergy or hypersensitivity to magnesium stearate, milk protein or the excipient lactose monohydrate, iodine, ipratropium bromide, tiotropium bromide, atropine and/or any of its derivatives.
* The subject has a significant clinical history of prostatic hypertrophy or narrow angle glaucoma.
* The subject has received an allogeneic bone marrow transplant.
* The subject has claustrophobia that may be aggravated by entering the whole body plethysmography cabinet.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
adverse events, vital signs,12-lead ECG, Holter and ECG monitoring,lung function and clinical lab tests. These will be taken pre-dose and at multiple time points up to 48h at each treatment period.

SECONDARY OUTCOMES:
- Plasma and urine concentrations of GSK704838 and derived pharmacokinetic parameters over 48h post-dose. - Serial sGaw, Raw and FEV1 measurements over 24h post-dose.
Serial specific airway conductance (sGaw), Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity measurements (FVC) over 24 hours post-dose of GSK704838 and tiotropium bromide.
Serial sGaw measurements over 48 hours for the last period in each cohort dose of GSK704838 and tiotropium bromide.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC6108697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register